CLINICAL TRIAL: NCT01618552
Title: Physician Training to Support Patient Self-Efficacy for Depression Care Behaviors
Brief Title: Training Doctors to Support Patient Self-Care of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012336397-1; R34MH095893 (NIH)
Record Dates: First submitted 2012-05-08; First posted 2012-06-13 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Depression; Diabetes
Keywords: Chronic disease; Cluster randomization; Comorbidity; Depression; Diabetes; Medical history taking; Office visits; Patient acceptance of health care; Patient compliance; Patient simulation; Physician patient relations; Primary health care; Randomized controlled trials; Self care; Self efficacy
MeSH Terms: conditions — Depression; Diabetes Mellitus; Chronic Disease; Patient Acceptance of Health Care; Patient Compliance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SEE IT training (interviewing skills) (Experimental): Intervention to train primary care physicians in the use of self-efficacy enhancing interviewing techniques (SEE IT) with patients who have coexisting depression and diabetes
  Interventions: Behavioral: SEE IT training
- Control (knowledge enhancement) (Active Comparator): Brief video clip designed to increase primary care physician awareness of new medication treatments for patients with diabetes
  Interventions: Other: Knowledge enhancement

INTERVENTIONS:
Behavioral: SEE IT training — Standardized patient instructors provide a scripted intervention to train primary care physicians in the use of self-efficacy enhancing interviewing techniques (SEE IT) during office visits with patients who have coexisting depression and diabetes
  Arms: SEE IT training (interviewing skills)
Other: Knowledge enhancement — Brief video clip designed to increase primary care physician awareness of new medication treatments for diabetes
  Arms: Control (knowledge enhancement)

SUMMARY:
This study will determine whether practicing primary care providers (PCPs) can be trained to support patient self-care of depression and co-existing diabetes during office visits, and begin to explore whether this might improve depression and diabetes outcomes, and whether the effects of the training generalize to patients with health conditions other than depression and diabetes. This is important because most patients with chronic conditions struggle with self-care and are seen in primary care, yet PCPs are seldom trained to support self-care.

DETAILED DESCRIPTION:
Many primary care patients struggle with health behaviors that can reduce depressive symptoms, such as adhering to prescribed treatments. Bolstering patient self-efficacy can improve health behaviors and outcomes, including those related to depression. However, current self-efficacy interventions are provided outside of primary care, and so cannot harness the power of therapeutic primary care provider (PCP)-patient relationships. Teaching PCPs to employ self-efficacy enhancing interviewing techniques (SEE IT) with patients would build upon existing therapeutic relationships, greatly increasing the reach of self-efficacy enhancement. The randomized controlled trial (RCT) in this proposal will examine whether, as compared with an attention control condition, a brief (< 1 hour) office-based intervention for practicing PCPs will lead to significantly greater use of SEE IT during unannounced follow-up SP encounters (postintervention and 3 months). The interventions will be delivered to PCPs during their regular office hours by standardized patient (SP) instructors. All study SPs will portray patients with both depression and diabetes, since these conditions commonly co-occur and entail a heavy burden of health-enhancing behaviors. Exploratory (due to limited statistical power) analyses will explore intervention effects on the following outcomes among real patients with co-occurring depression and diabetes: self-efficacy for depression and diabetes self-care, actual self-care behaviors (e.g. medication adherence), symptom severity, and health status. Further exploratory (due to limited statistical power) analyses will explore intervention effects on the following outcomes among real patients with various chronic conditions (ie, not limited to depression and diabetes): self-care self-efficacy, actual self-care behaviors, symptom severity, and health status. Pre- and post-RCT focus groups with stakeholders (PCPs, office staff, patients, and SP instructors) will guide refinement of the SEE IT intervention. The proposed research activities will inform the design (e.g. sample size) and conduct of a future R01-funded, multi-center, cluster RCT of the finalized intervention, adequately powered to examine effects on a range of patient outcomes; sustainability of effects on PCP interviewing over time; and generalizability to other practice settings and common co-morbid mental health and physical illness clusters. The SEE IT intervention begins to address the broader health needs of individuals with depression in primary care, and has unique potential to reduce the tremendous burden of mental illness related morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria: Physicians (targeted enrollment=56; actual enrollment=50)

* Currently in practice at a participating office within one of the 2 participating health systems (University of California Davis Primary Care Network, Sutter Sacramento Health System)
* Trained as a family physician, general practitioner, and/or general internist
* Able to read and speak English

Inclusion Criteria: Group of patients with diabetes and depressive symptoms (targeted enrollment=168; actual enrollment=15)

* Receive primary health care in one of the participating offices, from one of the participating primary care physicians
* Aged 18 years or older
* Able to read and speak English
* Self-report of adequate vision, hearing, and hand function to complete self-administered questionnaires on a touch screen notebook computer
* Have concurrent diagnoses of depression and diabetes, determined via medical record review
* Have at least mild depressive symptoms, manifested by a score of 10 or greater on a telephone-administered Patient Health Questionnaire (PHQ-9).
* Have an office visit scheduled with their assigned primary care provider within 1 month of study eligibility screening
* Made 2 or more of their primary care office visits during the preceding year with their assigned primary care provider

Inclusion Criteria: Group of patients with various health conditions, ie, not limited to diabetes and depression (targeted enrollment=336; actual enrollment=117)

* Receive primary health care in one of the participating offices, from one of the participating primary care physicians
* Aged 18 years or older
* Able to read and speak English
* Self-report of adequate vision, hearing, and hand function to complete self-administered questionnaires on a touch screen notebook computer
* Have an office visit scheduled with their assigned primary care provider within 1 month of study eligibility screening
* Made 2 or more of their primary care office visits during the preceding year with their assigned primary care provider

Exclusion Criteria: Patients (applies to all study patients)

* Self-report or medical record evidence of unstable overall medical status
* Self-report or medical record evidence of terminal illness
* Self-report or medical record evidence of bipolar disorder, chronic psychosis (schizophrenia or other), or personality disorder
* Self-report or medical record evidence of a history of attempted suicide
* Planned transfer of care to a health system other than the 2 participating systems within 6 months
* Inability to understand any of the screening questions, after appropriate explanation (e.g. due to cognitive impairment, developmental delay, or other reasons)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Physician use of self-efficacy enhancing interviewing techniques | During the 3 months after receiving intervention

SECONDARY OUTCOMES:
Patient self-efficacy for depression self-care | 5 minutes after an index visit with primary provider
Patient self-efficacy for diabetes self-care | 5 minutes after an index visit with primary provider
General self-care self-efficacy (all health conditions) | 5 minutes after an index visit with primary provider
Patient depressive symptoms | 3 months after an index visit with their primary care provider
Patient depression self-care behaviors | 3 months after an index visit with their primary care provider
Patient diabetes self-care behaviors | 3 months after an index visit with their primary care provider
Patient chronic illness self-care behaviors (generic) | 3 months after an index visit with their primary care provider
Patient adherence to depression and diabetes medications | 3 months after an index visit with their primary care provider
Patient adherence to chronic illness medications (generic) | 3 months after an index visit with their primary care provider
Patient adherence to depression counseling | 3 months after an index visit with their primary care provider
Patient mental health status | 3 months after an index visit with their primary care provider
Patient physical health status | 3 months after an index visit with their primary care provider
Patient glycemic control | 3 months after an index visit with their primary care provider
Wallston Multidimensional Health Locus of Control Scale | 5 minutes after an index visit with their primary care provider
  Perceived control over health
Healthcare Climate Questionnaire | 5 minutes after an index visit with their primary care provider
  Patient perception of degree to which primary care provider is autonomy supportive

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Jerant, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - Sutter Health Sacramento, Sacramento, California
  - University of California Davis Health System, Sacramento, California

REFERENCES:
- [Background] Jerant A, Kravitz RL, Azari R, White L, Garcia JA, Vierra H, Virata MC, Franks P. Training residents to employ self-efficacy-enhancing interviewing techniques: randomized controlled trial of a standardized patient intervention. J Gen Intern Med. 2009 May;24(5):606-13. doi: 10.1007/s11606-009-0946-4. Epub 2009 Mar 19. PMID 19296179
- [Derived] Jerant A, Kravitz RL, Tancredi D, Paterniti DA, White L, Baker-Nauman L, Evans-Dean D, Villarreal C, Ried L, Hudnut A, Franks P. Training Primary Care Physicians to Employ Self-Efficacy-Enhancing Interviewing Techniques: Randomized Controlled Trial of a Standardized Patient Intervention. J Gen Intern Med. 2016 Jul;31(7):716-22. doi: 10.1007/s11606-016-3644-z. Epub 2016 Mar 8. PMID 26956140